CLINICAL TRIAL: NCT01699490
Title: Role of Inflammation Factors and Insulin Resistance in the Pathophysiology and Treatment Response of Major Depressive Disorder
Brief Title: Role of Inflammation Factors and Insulin Resistance in Major Depressive Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Po-See, Chen, Associate Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSC 101-2314-B-006 -064 -MY3
Record Dates: First submitted 2012-09-30; First posted 2012-10-03 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Antidepressants; Insulin; Fluoxetine
MeSH Terms: conditions — Depressive Disorder, Major; Insulin Resistance | interventions — Fluoxetine; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoxetine + Valsartan (Experimental): The initial dose of fluoxetine was 20 mg once daily, which could be increased by 20 mg in divided doses to a maximal daily dose of 60 mg.
  Add-on treatment to 40 mg per day of valsartan
  Interventions: Drug: Fluoxetine + Valsartan
- Fluoxetine + Placebo (Active Comparator): The initial dose of fluoxetine was 20 mg once daily, which could be increased by 20 mg in divided doses to a maximal daily dose of 60 mg.
  Add-on treatment to placebo
  Interventions: Drug: Fluoxetine + Placebo

INTERVENTIONS:
Drug: Fluoxetine + Valsartan — The curative effect of fluoxetine add-on valsartan 40 mg per day for 12 weeks therapy in the treatment of major depressive disorder.
  Other Names: Prozac; Diovan
  Arms: Fluoxetine + Valsartan
Drug: Fluoxetine + Placebo — The curative effect of fluoxetine add-on placebo therapy in the treatment of major depressive disorder.
  Other Names: Prozac
  Arms: Fluoxetine + Placebo

SUMMARY:
The purpose of this study is to identify evidence-based guidelines for treating major depressive disorder to full remission in Taiwanese major depressive disorder (MDD) patients. To achieve this goal, the investigators aim to: (1) evaluate the risks and benefits of adjunctive pharmacotherapies for cognitive and metabolic consequences in MDD, and (2) clarify the shared biological mechanisms between mood, immune and metabolism homeostasis

DETAILED DESCRIPTION:
The prevalence of insulin resistance did not significantly differ among the healthy controls and drug-naïve MDD patients before and after antidepressant treatment. Meanwhile, the current study indicated that antidepressants might affect insulin secretion independently of the therapeutic effects on MDD. Therapeutic strategies considering both treatment effectiveness and glucose-insulin homeostasis in MDD patients are necessary.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16-65 years old
* Signed informed consent by patient or legal representative
* Hamilton Rating Scale for Depression (HDRS) scores ≥ 16
* A diagnosis of MDD according to DSM-IV criteria made by a specialist in psychiatry

Exclusion Criteria:

* Monoamine oxidase inhibitor or antidepressant treatment prior to entering the study
* A DSM-IV diagnosis of substance abuse within the past three months
* An organic mental disease, mental retardation or dementia
* A serious surgical condition or physical illness
* Patients who were pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | 12 weeks

SECONDARY OUTCOMES:
fasting plasma glucose | 12 weeks
fasting serum insulin | 12 weeks
C-reactive Protein, and IL-6 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Po See Chen, M.D., Ph.D, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- Department of Psychiatry, National Cheng-Kung University Hospital, Tainan, Taiwan